CLINICAL TRIAL: NCT07205081
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multi-Part, Single Ascending Dose and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ATTO-3712 in Healthy Adult Volunteers and Patients With Atopic Dermatitis
Brief Title: Safety, Tolerability and PK of ATTO-3712 in Healthy Volunteers and Patients With Atopic Dermatitis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Attovia Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATTO-3712-101
Record Dates: First submitted 2025-09-24; First posted 2025-10-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Normal Volunteers; Atopic Dermatitis (AD); Atopic Eczema; Atopic Eczema/Dermatitis (Non-Specific)
Keywords: Atopic Dermatitis; AD; Atopic Eczema; Ecema; Itch; Pruritus
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Pruritus

STUDY DESIGN:
Intervention Model Description: Single ascending dose, multiple ascending dose, randomized, double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ATTO-3712 single dose IV (Experimental): ATTO-3712 Dose level cohorts receiving a single dose IV
  Interventions: Drug: ATTO-3712
- Placebo single dose IV (Placebo Comparator): Placebo preparation to match Experimental Arm with single dose IV
  Interventions: Drug: Placebo
- ATTO-3712 single dose SC (Experimental): ATTO-3712 dose level cohorts receiving a single dose SC
  Interventions: Drug: ATTO-3712
- Placebo single dose SC (Placebo Comparator): Placebo preparation to match Experimental Arm with single dose SC
  Interventions: Drug: Placebo
- ATTO-3712 multiple dose SC (Experimental): ATTO-3712 administered to dose level cohorts in multiple SC doses
  Interventions: Drug: ATTO-3712
- Placebo multiple dose SC (Placebo Comparator): Placebo preparation to match Experimental Arm administered in multiple SC doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATTO-3712 — ATTO-3712
  Arms: ATTO-3712 multiple dose SC; ATTO-3712 single dose IV; ATTO-3712 single dose SC
Drug: Placebo — Placebo preparation to match ATTO-3712 dose
  Arms: Placebo multiple dose SC; Placebo single dose IV; Placebo single dose SC

SUMMARY:
The goal of this clinical trial is to assess the safety, tolerability, and pharmacokinetics of ATTO-3712 in healthy adults and patients with atopic dermatitis.

The main questions it aims to answer are:

What medical problems do participants have when taking ATTO-3712? How long does ATTO-3712 stay in the body after dosing? Researchers will compare ATTO-3712 to a placebo (a look-alike substance that contains no drug).

Participants will be dosed with ATTO-3712 or a placebo, visit the clinic for checkups and tests, and keep a diary of their symptoms.

DETAILED DESCRIPTION:
This is a 3-part study. Parts 1 and 2 will be a single and multiple ascending dose design, respectively, assessing the safety, tolerability, and PK of ATTO-3712 in healthy adult volunteers. Part 3 will consist of multiple doses in adult patients with atopic dermatitis to assess safety, tolerability, PK, and PD based on biomarkers in the blood.

ELIGIBILITY:
Parts 1&2 (Healthy Volunteers) Key Inclusion Criteria:

* Any sex or gender who is 18 to 65 years old, inclusive, at Screening.
* Body weight of 50 to 125 kg and body mass index (BMI) between 18.5 and 35 kg/m2
* Considered in good general health based on medical history, physical exam, 12-lead ECG, screening clinical laboratory findings, and vital signs
* Negative pregnancy test for participants of child-bearing potential.

Part 3 (Participants with Atopic Dermatitis) Key Inclusion Criteria:

* Any sex or gender who is 18 to 65 years old
* Body weight of 50 to 125 kg and BMI between 18.5 and 40 kg/m2
* Clinically confirmed diagnosis of active AD
* History of inadequate response to treatment with topical medications
* Baseline weekly mean of daily PP-NRS ≥ 4 at Day 1.
* EASI score of ≥ 16 at Screening and Day 1
* vIGA-AD score of ≥ 3 at Screening and Day 1
* ≥10% of body surface area (BSA) affected by AD at Screening and Day 1
* Use of topical bland emollient (moisturizer) at least once daily for at least 5 of the 7 days immediately before Day 1 and agrees to continue using that same emollient at the same frequency throughout the study
* Negative pregnancy test for participants of childbearing potential

Parts 1 & 2 (Healthy Volunteers) Key Exclusion Criteria

* Any clinically significant underlying illness
* History of malignancy within 5 years of Screening
* History of major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study
* History of uncontrolled asthma requiring rescue treatment with a bronchodilator for an increase in symptoms more than twice per week
* History of hypersensitivity (including anaphylaxis) to a biologic medication, vaccine, an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody), or to any of the IP excipients (sucrose, polysorbate 80, or histidine)
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or is positive for HIV
* Active or latent tuberculosis infection
* Smoking more than 20 cigarettes (or cigars, cigarillos, or e-cigarettes equivalent) per day
* History of drug or alcohol abuse
* Laboratory values outside of the normal range

Part 3 (Participants with Atopic Dermatitis) Key Exclusion Criteria:

* Any clinically significant underlying illness
* Presence of skin comorbidities that may interfere with study assessments
* Has taken prescription medication for the treatment of AD or other prohibited medication within the restricted time limits (defined in the protocol)
* Has applied topical corticosteroids within 2 weeks prior to dosing.
* History of malignancy within 5 years of Screening
* History of major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study
* History of uncontrolled asthma requiring rescue treatment with a bronchodilator for an increase in symptoms more than twice per week
* History of recurrent eczema herpeticum
* History of known primary immunodeficiency, is considered immunocompromised, history of untreated latent tuberculosis infection, has been treated for active tuberculosis in the past year, or has been treated for a parasitic infection in the past 6 months
* History of major depression
* History of hypersensitivity (including anaphylaxis) to a biologic medication, vaccine, an immunoglobulin product (plasma-derived or recombinant, eg, monoclonal antibody), or to any of the IP excipients (sucrose, polysorbate 80, or histidine)
* Participant has experienced significant flare(s) in AD in the 2 weeks prior to Screening or during the Screening period
* EASI score for the participant has more than doubled between Screening and Day 1
* Active HBV or HCV or is positive for HIV
* Participant is smoking more than 20 cigarettes (or cigars, cigarillos, or e-cigarettes equivalent to approximately 40 mg nicotine) per day
* Participant has an ECG with a QTcF > 450 msec for males or > 470 msec for females at Screening
* History of drug or alcohol abuse
* Laboratory values outside of the normal range

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of AEs | 0-113 Days for SAD; 0-143 Days for MAD
  The primary analysis will describe the incidence of AEs and laboratory abnormalities. AEs will be coded according to system organ class and preferred term using the Medical Dictionary for Regulatory Activities (MedDRA, version 28.0 or the current version). Their severity will be graded using the NCI CTCAE v5.0 or the current version.
Incidence of laboratory abnormalities | 0-113 Days for SAD; 0-143 days for MAD
  Clinical laboratory parameters (hematologic and blood chemistry) will be summarized by visit
Incidence of ECG abnormalities | 0-113 Days for SAD; 0-143 Days for MAD
  ECG findings (including QT abnormalities) will be summarized by visit.
Incidence of vital sign abnormalities | 0-113 Days for SAD; 0-143 Days for MAD
  Vital signs (systolic and diastolic blood pressure, temperature, heart rate) will be summarized by visit.

SECONDARY OUTCOMES:
Incidence of Anti-Drug Antibodies | 0-113 Days for SAD; 0-143 Days for MAD
  Baseline prevelance of ADA, changes in ADA status from prior to the first dose of IP to each applicable post-dose timepoint and ADA titer values for samples confirmed positive for ADA will be evaluated to assess the immunogenicity of single and multiple dose levels of ATT-3712.
Peak plasma concentration (Cmax) ATTO-3712 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include maximum concentration (Cmax) of ATTO-3712
Circulating half-life of ATTO-3712 (t1/2) | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include half-life (t1/2) of ATTO-3712.
Area Under the Plasma Concentration Versus Time Curve (AUC) | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include area under the plasma concentration-time curve (AUC).
Clearance Rate (C) of ATTO-3712 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include characterization of the clearance rate (C) of ATTO-3712.
Volume of Distribution (V) of ATTO-3712 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include characterization of the Volume of distribution (V) of ATTO-3712.
Bioavailability (F) of ATTO-3712 | 0-113 Days for SAD; 0-143 Days for MAD
  The pharmacokinetics of single and multiple dose levels of ATTO-3712 in participants will include characterization of the Bioavailability (F) of ATTO-3712.

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No